CLINICAL TRIAL: NCT07188935
Title: Effect of Glycemic Status on Antimicrobial Response in T2DM Patients With Recurrent UTI, Prospective Comparative Study
Brief Title: Glycemia and Antibiotic Efficacy in Diabetic Recurrent UTIs
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Al-Mustansiriyah University (Other)
Responsible Party: Principal Investigator, Maher Kadhum, Clinical Researcher, Al-Mustansiriyah University
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: MustansiriyahU ,80 ,3/m9/2024
Record Dates: First submitted 2025-09-01; First posted 2025-09-23 (Actual); Last update posted 2025-09-24 (Actual); Status verified 2025-09

CONDITIONS: T2DM (Type 2 Diabetes Mellitus)
MeSH Terms: conditions — Diabetes Mellitus, Type 2 | interventions — Ciprofloxacin; Tablets

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Non-diabetic patients with recurrent UTI (Active Comparator): Non diabetic patients with recurrent UTI receiving treatment
  Interventions: Drug: ciprofloxacin 500 mg tablet
- Diabetic patients with recurrent UTI (Other): Diabetic patients with recurrent UTI receiving treatments
  Interventions: Drug: ciprofloxacin 500 mg tablet

INTERVENTIONS:
Drug: ciprofloxacin 500 mg tablet — Administration of oral ciprofloxacin 500 mg twice daily for 7-14 days for the treatment of recurrent urinary tract infections in patients with type 2 diabetes mellitus, following local and international guidelines.

SUMMARY:
This study looked at how blood sugar control affects treatment of repeated urinary tract infections (UTIs) in people with type 2 diabetes. Ninety-nine patients at Al-Zahraa Teaching Hospital in Iraq were included. Some patients had good blood sugar control, while others did not. All were treated with antibiotics, and doctors checked if the infection was cured after 14 days and if it came back within 30 days. The study helps show how diabetes management can affect recovery from UTIs and the chance of infection returning.

DETAILED DESCRIPTION:
Recurrent urinary tract infections (rUTIs) are a frequent complication among patients with type 2 diabetes mellitus (T2DM), associated with impaired immune function, glycosuria, and increased risk of antimicrobial resistance. While UTIs are common in both diabetic and non-diabetic patients, recurrence rates and treatment failures are higher in T2DM. Few prospective studies have evaluated the effect of glycemic control on antimicrobial response in this population.

This prospective comparative study enrolled 99 patients with recurrent UTIs, including 58 with T2DM, at Al-Zahraa Teaching Hospital, Wasit Province, Iraq. Patients with diabetes were stratified into groups based on glycemic control (good vs. poor). Antimicrobial therapy was administered according to hospital guidelines, and treatment response was evaluated after 14 days (clinical cure). Patients were followed for 30 days to monitor recurrence.

The primary objective was to assess whether glycemic status influences antimicrobial treatment outcomes in patients with rUTIs. Secondary objectives included evaluating recurrence rates and identifying potential risk factors for treatment failure. Findings from this study highlight the importance of optimizing glycemic control as part of the overall management of recurrent UTIs in patients with T2DM.

ELIGIBILITY:
Inclusion Criteria:

* Patients age >18 years, both sex
* Patient with known history of T2DM at least 1 year
* Patients diagnosed with rUTI according to the positive GUE as in practice guideline
* Patients with different glycemic status according to the HbA1c level, and on different treatment for T2DM accordingly.
* Patients with non-diabetic rUTI as active comparator.
* Patients who had the ability to communicate to answer study questionnaire.

Exclusion criteria:

* Type 1 diabetic patients on insulin therapy were excluded.
* T2DM Patients who were using Sodium-glucose co-transporter-2 inhibitors (SGLT-2) (because of their renal -related side effect).
* Patients who received any antimicrobial treatment within the last 72 hours of their enrollment.
* Women patients with recurrent vaginitis or urinary incontinence.
* Men patients with BPH or over flow incontinence ( as a cause for r UTI).
* Patients with chronic disease other than T2DM that may cause rUTI ( eg. CKD, Spinal cord injury. kidney stone).
* Pregnancy and lactation

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 99 (Actual)
Dates: Start 2024-10-30 (Actual); Primary Completion 2025-06-20 (Actual); Study Completion 2025-06-20 (Actual)

PRIMARY OUTCOMES:
treatment success will be defined as simultaneous absence of symptoms and GUE showing <5 pus cells/HPF and MARS-10 score ≥8. Unit of measure: % of participants meeting all criteria. | Up to 14 days after completion of antimicrobial therapy
treatment success will be defined as simultaneous absence of symptoms and GUE showing <5 pus cells/HPF after 30 days of treatment initiation | Day 30 after treatment initiation

CONTACTS AND LOCATIONS:
Locations (1):
- Al-Zahraa Teaching Hospital, Wasit, Iraq, Kut, Wasit Governorate, Iraq

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- See also: Related Info — https://doi.org/10.1016/0163-4453(92)92876-K
- Available data/document: Individual Participant Data Set: rUTI_T2DM_2025 — https://doi.org/10.1016/0163-4453(92)92876-K — De-identified participant-level data, including demographics, glycemic status, UTI recurrence, antimicrobial therapy, adherence (MARS), and clinical outcomes. Available upon request for research purposes.